CLINICAL TRIAL: NCT00214682
Title: Beyond Ageing Project: A RCT to Assess the Benefit of Improving Mental Health Literacy as Well as the Effect of Folate and B12, and Physical Activity, in Preventing Major Depression and Cognitive Decline Among Older Australians
Brief Title: Beyond Ageing Project: A Study for the Prevention of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian National University (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); University of Sydney (Other); Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Responsible Party: Principal Investigator, Dr Janine Walker, Research Fellow, Australian National University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2004/188 HREC; 2005/483 (TGA)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Depression; Depressive Disorder
Keywords: Depression; Cognition; Depressive disorder; Mental health literacy; Older adults; Randomzed controlled trial
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Folic acid (400mcg) + Vitamin B12 (100 mcg) (Experimental): The vitamin intervention was a daily oral dose of one tablet consisting of folic acid 400 mcg + vitamin B12 100 mcg. The folic acid dose of 400 mcg / day was selected as it has been shown to be the dose associated with 90% of the maximal decrease in plasma homocysteine concentration for older individuals. Participants received 1 bottle x 200 tablets in six-month supplies at baseline, 6 months, 12 months, and 18 months. Adherence was monitored by telephone interviews (6 weeks, 6-, 12-, and 24 months) and 10 brief telephone tracking calls (1 - 5 weeks, and 4-, 8-, 13-, 18-, and 22-months).
  Interventions: Drug: Folate (400mcg) and Vitamin B12 (100 mcg)
- Mediated physical activity promotion (Experimental): Individuals in the Physical Activity Promotion group received a manual designed to promote older individuals' physical activity participation to the level recommended to gain both physical and mental health benefits. The framework of the physical activity manual was informed by social cognitive theory and the transtheoretical model, and comprised five sections that reflect stages of behaviour change, including; precontemplation, contemplation, preparation, action, and maintenance. The manual contained evidence-based strategies and skills to assist people in increasing their physical activity levels. Participants received a pedometer at the commencement of the intervention as pedometry step / minute values are useful as an indicator of moderate to vigorous physical activity with total number of steps for one week recorded during the brief telephone calls at 1-5 weeks, and 4-, 8-, 13-, 18-, and 22- months.
  Interventions: Behavioral: mediated physical activity promotion
- Mental health literacy (Experimental): This MHL intervention comprised 10 modules, with nine of these specifically written for older adults. Modules 1 to 5 comprised information on depression and the evidence-based treatment for older adults. The additional MHL modules were booklets addressing evidence-based strategies and treatments for depression. It was delivered in a way to foster support and ensure that participants worked through the material systematically. Modules 1 to 5 were delivered in consecutive weeks as previous research indicates that the maximum impact of MHL on depressive symptoms may occur within the first six weeks of the intervention. Telephone interviewers contacted participants once a week for 5 consecutive weeks to motivate and support participants. There were an additional 5 check-in telephone calls, and Modules 6 to 10 of the MHL material that were delivered via postal mail at 4- (Module 6), 8- (Module 7), 13- (Module 8), 18- (Module 9), and 22- months (Module 10).
  Interventions: Behavioral: Mental health literacy
- Placebo tablet (Placebo Comparator): A placebo tablet was the attention control intervention for the folic acid + vitamin B12 intervention group. Participants received 1 bottle x 200 tablets in 6-month supplies at baseline, 6 months, 12 months, and 18 months. Adherence was monitored by telephone interviews (6 weeks, 6-, 12-, and 24 months) and 10 brief telephone tracking calls (1 - 5 weeks, and 4-, 8-, 13-, 18-, and 22-months) during which participants counted their left-over tablets.
  Interventions: Drug: placebo
- Nutrition information (Active Comparator): The attention control intervention for the physical activity intervention was printed nutrition literacy and included information concerning the recommended dietary guidelines for older Australians, as well as strategies and additional information to facilitate beneficial dietary behaviours. The same procedure was adhered to as the physical activity intervention to ensure adequate attention control. Participants in the nutrition promotion intervention received 5 brief telephone calls from an interviewer to facilitate adherence to the intervention, and to offer support and clarification of the materials. Participants received five further brief telephone calls as well as nutrition newsletters that were delivered via postal mail at 4-, 8-, 13-, 18-, and 22- months.
  Interventions: Behavioral: Nutrition information
- Pain and arthritis management information (Active Comparator): Pain and Arthritis Information was used as the attention control intervention for the MHL intervention and comprised 10 modules. Modules 1 to 5 were contained in an Arthritis Australia consumer guide for arthritis management. Modules 6 to 10 were a series of information pamphlets on pain management, osteoporosis and falls prevention. The delivery of the Pain Information was identical to the MHL intervention with Modules 1 to 5 distributed via postal mail in five consecutive weeks (1-5 weeks), while the remaining intervention modules were delivered at 4- (Module 6), 8- (Module 7), 13- (Module 8), 18- (Module 9), and 22- months (Module 10). Participants also received 10 brief calls from a telephone interviewer that coincided with receiving the print intervention materials.
  Interventions: Behavioral: pain and arthritis management information

INTERVENTIONS:
Drug: Folate (400mcg) and Vitamin B12 (100 mcg) — The vitamin intervention was a daily oral dose of one tablet consisting of folic acid 400 mcg + vitamin B12 100 mcg. The folic acid dose of 400 mcg / day was selected as it has been shown to be the dose associated with 90% of the maximal decrease in plasma homocysteine concentration for older individuals. Participants received 1 bottle x 200 tablets in six-month supplies at baseline, 6 months, 12 months, and 18 months. Adherence was monitored by telephone interviews (6 weeks, 6-, 12-, and 24 months) and 10 brief telephone tracking calls (1 - 5 weeks, and 4-, 8-, 13-, 18-, and 22-months).
  Arms: Folic acid (400mcg) + Vitamin B12 (100 mcg)
Behavioral: mediated physical activity promotion — Individuals in the Physical Activity Promotion group received a manual designed to promote older individuals' physical activity participation to the level recommended to gain both physical and mental health benefits. The framework of the physical activity manual was informed by social cognitive theory and the transtheoretical model, and comprised five sections that reflect stages of behaviour change, including; precontemplation, contemplation, preparation, action, and maintenance. The manual contained evidence-based strategies and skills to assist people in increasing their physical activity levels. Participants received a pedometer at the commencement of the intervention as pedometry step / minute values are useful as an indicator of moderate to vigorous physical activity with total number of steps for one week recorded during the brief telephone calls at 1-5 weeks, and 4-, 8-, 13-, 18-, and 22- months.
  Arms: Mediated physical activity promotion
Behavioral: Mental health literacy — Comprises 10 modules, with nine of these specifically written for older adults. Modules 1 to 5 comprised information on depression and the evidence-based treatment for older adults. The additional MHL modules were booklets addressing evidence-based strategies and treatments for depression. It was delivered in a way to foster support and ensure that participants worked through the material systematically. Modules 1 to 5 were delivered in consecutive weeks as previous research indicates that the maximum impact of MHL on depressive symptoms may occur within the first six weeks of the intervention. Telephone interviewers contacted participants once a week for 5 consecutive weeks to motivate and support participants. There were an additional 5 check-in telephone calls, and Modules 6 to 10 of the MHL material that were delivered via postal mail at 4- (Module 6), 8- (Module 7), 13- (Module 8), 18- (Module 9), and 22- months (Module 10).
  Arms: Mental health literacy
Drug: placebo — A placebo tablet was the attention control intervention for the folic acid + vitamin B12 intervention group. Participants received 1 bottle x 200 tablets in 6-month supplies at baseline, 6 months, 12 months, and 18 months. Adherence was monitored by telephone interviews (6 weeks, 6-, 12-, and 24 months) and 10 brief telephone tracking calls (1 - 5 weeks, and 4-, 8-, 13-, 18-, and 22-months) during which participants counted their left-over tablets.
  Other Names: placebo tablet
  Arms: Placebo tablet
Behavioral: Nutrition information — The attention control intervention for the physical activity intervention was printed nutrition literacy and included information concerning the recommended dietary guidelines for older Australians, as well as strategies and additional information to facilitate beneficial dietary behaviours. The same procedure was adhered to as the physical activity intervention to ensure adequate attention control. Participants in the nutrition promotion intervention received 5 brief telephone calls from an interviewer to facilitate adherence to the intervention, and to offer support and clarification of the materials. Participants received five further brief telephone calls as well as nutrition newsletters that were delivered via postal mail at 4-, 8-, 13-, 18-, and 22- months.
  Arms: Nutrition information
Behavioral: pain and arthritis management information — Pain and Arthritis Information was used as the attention control intervention for the MHL intervention and comprised 10 modules. Modules 1 to 5 were contained in an Arthritis Australia consumer guide for arthritis management. Modules 6 to 10 were a series of information pamphlets on pain management, osteoporosis and falls prevention. The delivery of the Pain Information was identical to the MHL intervention with Modules 1 to 5 distributed via postal mail in five consecutive weeks (1-5 weeks), while the remaining intervention modules were delivered at 4- (Module 6), 8- (Module 7), 13- (Module 8), 18- (Module 9), and 22- months (Module 10). Participants also received 10 brief calls from a telephone interviewer that coincided with receiving the print intervention materials.
  Arms: Pain and arthritis management information

SUMMARY:
The purpose of this study is to determine whether folate and vitamin B12, physical activity and mental health literacy can prevent depression, and folate and vitamin B12 and physical activity can prevent cognitive impairment in older people. Also the study aims to assess the benefits for older people in improving their knowledge about mental health in relation to depression.

DETAILED DESCRIPTION:
While preventive efforts for depression have tended to focus on adolescent and young adult populations, other stages of the lifespan also provide opportunities for prevention. With older people, there are certain risk and aetiological factors, which become more prominent and require preventive action at that point in the lifespan. The aim of this study is to determine the efficacy of various interventions in preventing depression and cognitive decline among older people who are at high risk of developing major depression because they are currently suffering from depressive symptoms.

The study has three interventions; i) folate and vitamin B12, ii) physical activity; and iii) mental health literacy. Participants will be randomly allocated to receive each combination of the interventions (folate and vitamin B12 or placebo, physical activity intervention programme or physical activity no-intervention control, mental health literacy intervention [containing written modules with information about depression that is relevant to older people] or mental health literacy no-intervention control group). Participants will receive these interventions over a two-year period with regular assessments across that time period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-74 years with some depressive symptoms, assessed using the Kessler 10 Psychological Distress Scale [K10] (Andrews & Slade, 2001)

Exclusion Criteria:

Any of the following:

* Those currently taking medication or receiving psychological treatment for depression
* A report of a medical diagnosis of bipolar disorder/mania
* History of epilepsy
* Diagnosed with cancer and/or on antifolate therapy
* Have a diagnosis of dementia or Alzheimer's disease
* Are currently taking vitamin supplements containing folate, B2, B6 or B12 at a dose exceeding 25% of the recommended daily intake.
* Medical contradictions to exercise (e.g., significant orthopaedic problems or cardiovascular disease that would prevent regular aerobic exercise)
* Ongoing participation in regular aerobic exercise.

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 909 (Actual)
Dates: Start 2005-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline, 6 weeks, 6-, 12-, 48-, and 51 month followups.
  The Patient Health Questionnaire - 9 (PHQ - 9) is a brief self-administered diagnostic instrument for depressive symptoms with items derived from the nine diagnostic criteria for Major Depression Disorder using the DSM - IV. The items are coded "0" (not at all) to "3" (nearly every day) for the most recent 2-week period, with possible scores ranging from 0 to 27, higher scores indicating greater depression severity. The PHQ - 9 is used in research and clinical settings, and can be administered via telephone. Studies support its reliability, validity, and ability to detect change over time.

SECONDARY OUTCOMES:
Physical activity level | Baseline, 6 weeks, 6-, 12-, 48-, and 51 month followups.
  The International Physical Activity Questionnaire - Short Form (IPAQ - SF) was used as a self-report measure of physical activity. The purpose of the IPAQ is to survey physical activity in large groups or populations. The IPAQ allows for a total of metabolic equivalent (MET) units expended in the most recent seven-day period.
Cognitive impairment | Baseline, 12-, and 48-month followups.
  The modified Telephone Interview of Cognitive Status has a max. total score= 39, and comprises 4 domains: orientation; recent memory and delayed recall; attention; and, semantic memory. It has excellent discrimination in cognitive performance in the general population. Processing speed was measured (Brief Test of Adult Cognition-Telephone) with the task to count backwards quickly from 100 by 1's for 30 seconds The Informant Questionnaire on Cognitive Decline in the Elderly was given at 2yr FU to a person who had known the participant for > 2yrs. It measures cognitive decline and dementia.
Physical health outcomes | Baseline, 6-week, 6-, 12-, 24-, and 48-month followups.
  A health checklist was given to determine current health status with items addressing the following health domains: cardiovascular, pulmonary, musculoskeletal, psychiatric, vision, and renal health; cancer, diabetes, and epilepsy. Blood collections were also used at baseline, 12- and 24 months to further investigate health including: thyroid stimulating hormone; liver and kidney function; fasting cholesterol and blood glucose; C-reactive protein; and haematological parameters.
B12 levels | Baseline, 12-, and 48-month followups.
  Serum vitamin B12 was measured using chemiluminscent microparticle assays (Architect i2000, Abbott Laboratories). This allowed a check on whether participants were taking the supplements, and to initially to comply with inclusion/exclusion criteria.
Folate status | Baseline, 12-, and 48-month followups.
  Red cell folate was measured using chemiluminscent microparticle assays (Architect i2000, Abbott Laboratories). This allowed a check on whether participants were taking the supplements, and as part of the initial screening process to comply with our inclusion/exclusion criteria.
Homocysteine | Baseline, 12- and 24-month followups.
  A fluorescence polarization immunoassay was used for the quantitative determination of total L-homocysteine in plasma (AxSYM, Abbott Laboratories). This allowed us to establish any changes in Hcy concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Helen Christensen, PhD, Principal Investigator — Centre for Mental Health Research, ANU; Professor Anthony F Jorm, PhD, Principal Investigator — ORYGEN Research Centre, University of Melbourne; Professor Ian Hickie, PhD, Principal Investigator — Brain and Mind Research Institute, University of Sydney; Dr Janine G Walker, PhD, Principal Investigator — Centre for Mental Health Research, Australian National University, Canberra, Australia
Locations (1):
- Australian National University, Canberra, Australian Capital Territory, Australia

REFERENCES:
- [Derived] Walker JG, Batterham PJ, Mackinnon AJ, Jorm AF, Hickie I, Fenech M, Kljakovic M, Crisp D, Christensen H. Oral folic acid and vitamin B-12 supplementation to prevent cognitive decline in community-dwelling older adults with depressive symptoms--the Beyond Ageing Project: a randomized controlled trial. Am J Clin Nutr. 2012 Jan;95(1):194-203. doi: 10.3945/ajcn.110.007799. Epub 2011 Dec 14. PMID 22170358
- [Derived] Christensen H, Aiken A, Batterham PJ, Walker J, Mackinnon AJ, Fenech M, Hickie IB. No clear potentiation of antidepressant medication effects by folic acid+vitamin B12 in a large community sample. J Affect Disord. 2011 Apr;130(1-2):37-45. doi: 10.1016/j.jad.2010.07.029. PMID 20805005
- [Derived] Walker JG, Mackinnon AJ, Batterham P, Jorm AF, Hickie I, McCarthy A, Fenech M, Christensen H. Mental health literacy, folic acid and vitamin B12, and physical activity for the prevention of depression in older adults: randomised controlled trial. Br J Psychiatry. 2010 Jul;197(1):45-54. doi: 10.1192/bjp.bp.109.075291. PMID 20592433